CLINICAL TRIAL: NCT06965283
Title: The Effect of Integrating Postpartum Family Planning Intervention With Maternal & Child Health Services on Modern Postpartum Contraceptive Use and Service Improvement in Northeast Ethiopia
Brief Title: The Effect of Integrating Postpartum Family Planning Intervention With Maternal & Child Health Services
Acronym: PPFP MCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jimma University (Other)
Collaborators: Wollo University (Other)
Responsible Party: Principal Investigator, Delelegn Tsegaye, Principal investigator, Jimma University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: JUIH/IRB/0474/25; Jimma UNiversity (Other: Jimma University)
Record Dates: First submitted 2025-04-11; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Postpartum Family Planning; Modern Contraceptive Use
Keywords: Modern contraceptive use; Postpartum family planning; Service integration; Maternal & child health services

STUDY DESIGN:
Intervention Model Description: All postpartum mothers who come to the hospital for labor/delivery, infant immunization, PMTCT (Prevention of Mother-to-Child Transmission), postnatal care (PNC), or under-five childcare services will be screened and counseled for postpartum family planning (PPFP). Those who decide to use a modern contraceptive method will either be referred to family planning units or provided with their chosen method directly.
  Postpartum mothers who do not initially decide to use a modern contraceptive method will receive additional counseling during their next visit. The intervention will be implemented by nurses and midwives working in selected maternal and child health units. These healthcare providers will receive a three-day PPFP training session delivered by a senior obstetrician-gynecologist, public health expert, and maternal/reproductive health specialist, all of whom are certified Training of Trainers. Coaching and mentoring will also be provided to ensure they acquire adequate knowledge.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- This arm will be given the multiple behaviour change intervention (Active Comparator): The intervention package includes:
  1. PPFP refresher training for maternal and child health (MCH) providers across all MCH units (labor/delivery, postnatal care [PNC], immunization, PMTCT [Prevention of Mother-to-Child Transmission], and under-five childcare clinics).
  2. Weekly mentoring (internal and external) led by senior gynecologists, obstetricians, and midwives at intervention hospitals. Mentoring sessions use anatomical models to address knowledge and skill gaps. MCH service coordinators also participate in training sessions to facilitate coaching and monitoring.
  3. Standardized training modules based on guidelines developed by the Ethiopian Ministry of Health.
  4. Monthly supportive supervision of PPFP services, conducted jointly by MCH unit coordinators and hospital management teams. This ensures early identification of bottlenecks and prompt resolution of challenges.
  5. Monitoring of contraceptive methods and other materials availability
  Interventions: Behavioral: Providing training and Mentoring
- The non intervention group were not given the intervention. Standard care will be continued (No Intervention): Usual care can be continued. No intervention can be given

INTERVENTIONS:
Behavioral: Providing training and Mentoring — The intervention packages are providing postpartum family planning training at each MCH units, Using WHO PPFP counseling toolkit, mentoring health care provider to fill knowledge and skill gap, contraceptive logistic availability, and regular supportive supervision
  Arms: This arm will be given the multiple behaviour change intervention

SUMMARY:
This study aims to explore the effectiveness of integrated package interventions within maternal and child health services in improving modern postpartum contraceptive use in northeast Ethiopia. Its primary objective is to enhance the utilization of postpartum contraceptive methods to reduce unmet needs for these methods in the Amhara region of Ethiopia.

DETAILED DESCRIPTION:
One of the advantages of this intervention study is that the provision of postpartum family planning (PPFP) services will not be limited to a few points of contact but will instead be integrated into the entire maternal care continuum. However, many studies in other countries have not used quasi-experimental or intervention study designs.

This pre/post-test interventional study with a control group employs extended observation and intervention periods, along with repeated measurements at the aggregate/population level. This approach will better capture changes in postpartum family planning (PPFP) integration and the factors influencing the use of integrated PPFP services.

This dissertation research project will contribute to various stakeholders. For health professionals and managers, it will enhance their knowledge and skills regarding the impact of integrating PPFP with maternal health services and its role in improving maternal and child health. It will also identify facilitators and barriers to PPFP integration with maternal and child health services.

Healthcare providers will gain leadership and communication skills in client-centered counseling and its effect on postpartum contraceptive use. The study highlights the importance of provider-led PPFP counseling and interventions for postpartum mothers visiting health facilities for maternal and child care services.

Reproductive-age mothers will benefit from this study by gaining access to modern contraceptives immediately after childbirth and up to 12 months postpartum. This will improve their health and their children's well-being by enabling them to space or limit births as desired. PPFP use, as shown in prior studies, significantly reduces maternal and neonatal morbidity and mortality by preventing unintended pregnancies.

Donors and non-governmental organizations (NGOs) can use these findings to strengthen healthcare systems through targeted support, including regular mentoring, logistics, and capacity-building training for providers and management teams.

Researchers will benefit from this study's findings as a baseline for future research, leveraging its recommendations and addressing its limitations. The project aims to assess the effect of integrating PPFP with maternal and child health services (e.g., postnatal care, delivery, PMTCT, immunization, and under-five childcare) and to identify the level of integration, facilitators, and barriers.

Policymakers, the Ethiopian Ministry of Health, and regional health bureaus can use these findings to design strategies aligned with the Sustainable Development Goals (SDGs), particularly reducing unmet PPFP needs. One SDG targets improved maternal health through integrated maternal and child health services, which this study supports by promoting PPFP use and advancing maternal and neonatal health outcomes.

ELIGIBILITY:
Inclusion criteria

* Postpartum mothers who gave birth one year preceding the survey
* All postpartum mothers who come for maternal and child health services(PMTCT, PNC, labor, delivery, under 5 OPD care and immunization services and post-partum women units)
* Those mothers whose age are between 18- 49 years old Exclusion criteria

  * Those participants who were seriously ill
  * Mentally unable to communicate

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 607 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Modern postpartum contraceptive use | Up to six months
  The primary outcome measure is modern postpartum contraceptive use, assessed via interviewer-administered questionnaires. Data were collected using standardized, pre-tested tools by trained midwives with prior data collection experience.
  Quantitative data will be analyzed using STATA 17 software with a Generalized Estimating Equation (GEE) model. The outcome variable was evaluated by measuring the effectiveness of the intervention package, which was delivered by trained healthcare providers across selected maternal and child health (MCH) units. These units included labor/delivery, immunization, postnatal care (PNC), PMTCT (Prevention of Mother-to-Child Transmission), and under-five child outpatient services.
  The study followed a pre/post-intervention design: a baseline assessment was conducted first, followed by a six-month intervention period, and a post-intervention assessment. The intervention's effect will be evaluated using difference-in-differences analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Gurmesa Tura Professor, PhD, Study Director — Jimma University; Sisay Eshete Assistant professor, Msc, Study Chair — Wollo University; Getabalew Tsegaye Mr., Bsc, Study Director — Unaffilated
Locations (2):
- Ethiopia (2):
  - Dessie Comprehensive specialized Hospital, Dessie, Amhara
  - Dessie referral Hospital, Dessie, Amhara

IPD SHARING:
Plan to Share IPD: No
The result of this study will be published at reputable journal. So the data can be accessed in the published paper.

REFERENCES:
- See also: It showed on postpartum family planning integration and its effect on modern contraceptive use — https://www.joghr.org/article/13511-effect-of-integrating-postpartum-family-planning-into-the-health-extension-program-in-ethiopia-on-postpartum-adoption-of-modern-contraception/stats